CLINICAL TRIAL: NCT01428440
Title: A Positron Emission Tomography (PET) Study to Evaluate 18FML10 as an Imaging Agent for Tumour Apoptosis
Brief Title: PET Study to Study Tumour Apoptosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early as the results did not support study objectives and were not as significant as expected.
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 113236
Record Dates: First submitted 2011-08-25; First posted 2011-09-05 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- no treatment (Other)
  Interventions: Radiation: 18FML10

INTERVENTIONS:
Radiation: 18FML10 — apoptosis imaging radio ligand

SUMMARY:
Apoptosis or programmed cell death is disrupted in cancer cells allowing them to live longer. A number of anti-cancer agents induce apoptosis as a mechanism of drug action to get rid of cancers. A biomarker that would allow apoptosis in tumours to be imaged directly would provide a powerful new tool for oncology drug development and potentially contribute to improved patient care. In this study, we propose to evaluate [18F]ML10-PET for imaging tumour apoptosis in patients receiving standard chemotherapy treatment for their cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients >18 years of age at screening with histological or cytological diagnosis of non-Hodgkin's lymphoma, small cell lung cancer, breast or ovarian cancer who have been worked up clinically (see below) and due to receive standard chemotherapy treatment, but enrolled prior to the initiation of chemotherapy.
* A female subject is eligible to participate if she is of non-childbearing potential or if she is of childbearing potential and agrees to use one of the contraception methods listed. Male subjects are eligible to participate if he also agrees to use one of the contraception methods listed.
* Tumour that is considered by the investigator to be able to be imaged using PET (about 2cm in size or more)
* Able to lie comfortably on back for up to 65 minutes at a time.
* Capable of giving written informed consent, and willing and able to comply with the requirements and restrictions listed in the consent form.
* Patients deemed to be fit to receive chemotherapy treatment by their oncologist.
* WHO performance status 0, 1 or 2.

Exclusion Criteria:

* Any medical or psychiatric diagnoses or symptoms or social situations that in the view of the investigator would limit compliance with study requirements.
* Pregnant or breast feeding females.
* Received any other anticancer therapy (radiotherapy, chemotherapy, or immunotherapy) or any other investigational agent, including an investigational anti-cancer agent within 28 days prior to the first [18F]ML10-PET scan.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Inability to comply with contraceptive guidelines during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Apoptosis imaging | 2.5 years
  Evaluate feasibility of apoptosis imaging with [18F]ML10 PET/CT in

SECONDARY OUTCOMES:
[18F]ML10 tumour uptake | 2.5 years
  To explore the relationship between [18F]ML10 tumour uptake and tissue markers
Image optimisation time | 2.5 years
  To identify an optimal image acquisition time relative to treatment
Develop Imaging protocols | 2.5 years
  To develop simplified imaging protocols for future drug development studies
serum markers | 2.5 years
  To explore the potential role of serum markers in relation to imaging
Oncology patients | 2.5 years
  To evaluate oncology patient compliance and attitudes to imaging studies

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, London, London
  - GSK Investigational Site, London